CLINICAL TRIAL: NCT02041520
Title: Effect of Omega 3 Fatty Acids on Oxidative Stress in Seropositive HIV Patients
Brief Title: Effect of Omega 3 Fatty Acids on Oxidative Stress in HIV Seropositive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, Norma Amador Licona, PhD, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: R-2011-785-058
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-07

CONDITIONS: HIV/AIDS
Keywords: Seropositive HIV; Omega 3 fatty acids; Oxidative stress
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Fatty Acids, Omega-3; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega 3 fatty acids (Experimental): omega 3 fatty acids, 2.4 g per day, requiring intake 2 capsules (600mg each one) in the morning and two at night (Zonelabs, Marblehead MA) for 6 months.
  Interventions: Drug: omega 3 fatty acids
- Placebo (Placebo Comparator): Placebo (olive oil gelcaps) in similar presentation as omega 3 fatty acids, requiring intake 2 capsules in the morning and two at night (Perfect Source, Fullerton CA, product code number PER 1016, lot number 8A0019/1600-1)
  Interventions: Other: placebo

INTERVENTIONS:
Drug: omega 3 fatty acids — omega 3 fatty acids will be administered until progression or unacceptable toxicity develops during 6 months follow up.
  Other Names: Zonelabs, Marblehead MA
  Arms: Omega 3 fatty acids
Other: placebo — olive oil in similar presentation of omega 3 fatty acids will be administered until progression or unacceptable toxicity develops during 6 months follow up.
  Other Names: olive oil
  Arms: Placebo

SUMMARY:
Introduction: Highly active antiretroviral therapy (HAART) has showed its effectiveness in the prevention of complications in seropositive for HIV patients. However, they develop some manifestations such as lipodystrophy, dyslipidemia, and glucose intolerance increasing cardiovascular risk.

Clinical trials in general population and in patients on hemodialysis have demonstrated a significant reduction in cardiovascular events using fish oil. Omega-3 fatty acids are believed to be beneficial in prevention of atherosclerosis reducing lipids levels specially triglycerides. Also in general populations it has been described a benefit effect of omega 3 acids on oxidative stress.

Objective: to know the effect of omega 3 acids on different markers of oxidative stress in seropositive HIV patients.

Methods: We will perform a randomized parallel controlled clinical trial in seropositive HIV patients from 20 to 55 years old on clinical score A1, A2, B1 or B2 who received HAART. They will be randomly assigned to receive omega 3 fatty acids 2.4 g (Zonelabs, Marblehead MA) or placebo for 6 months. At baseline anthropometric measurements, lipid profile, glucose and stress oxidative levels (nitric oxide, malondialdehyde, total glutathion, and lipid peroxidation products) will be evaluated.

Sample size was calculated according to different variables. We selected the biggest one calculated for a difference in nitric oxide of 25% after treatment between groups and a standard deviation (SD) value of 10µmol/L. Whit this information we obtained a sample size of 31 patients per group for an 80% statistical power with α= 0.05. Assuming a 15% patient lost, a sample size of 35 per group was considered.

ELIGIBILITY:
Inclusion Criteria:

* Seropositive HIV patients from 20 to 55 years old
* On clinical score A1, A2, B1 or B2
* Patients who received highly active antiretroviral therapy for at least 3 months.

Exclusion Criteria:

* Patients diagnosed with diabetes mellitus
* Patients diagnosed with hypertension
* Patients using hypolipidemic agents or diagnosed with dyslipidemia before receiving HAART therapy.
* Patients using protease inhibitors

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-01; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norma Amador, PhD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, León, Guanajuato, Mexico

REFERENCES:
- [Derived] Amador-Licona N, Diaz-Murillo TA, Gabriel-Ortiz G, Pacheco-Moises FP, Pereyra-Nobara TA, Guizar-Mendoza JM, Barbosa-Sabanero G, Orozco-Avina G, Moreno-Martinez SC, Luna-Montalban R, Vazquez-Valls E. Omega 3 Fatty Acids Supplementation and Oxidative Stress in HIV-Seropositive Patients. A Clinical Trial. PLoS One. 2016 Mar 25;11(3):e0151637. doi: 10.1371/journal.pone.0151637. eCollection 2016. PMID 27015634

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (olive oil gelcaps) in similar presentation as omega 3 fatty acids, requiring intake 2 capsules in the morning and two at night (Perfect Source, Fullerton CA, product code number PER 1016, lot number 8A0019/1600-1)
  omega 3 fatty acids: omega 3 fatty acids will be administered until progression or unacceptable toxicity develops during 6 months follow up.
Period: Overall Study
Arm/Group | Omega 3 Fatty Acids | Placebo
Started | 35 (35 patients randomly assigned to omega 3 fatty acids) | 35 (35 patients randomly assigned to placebo)
Completed | 29 | 28
Not Completed | 6 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Hypothiroidism identified during follow- | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega 3 Fatty Acids | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (9.5) | 39.9 (8.0) | 39.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 28 | 23 | 51
Region of Enrollment [Number; unit: participants]
  Mexico | 35 | 35 | 70
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (4.3) | 26.5 (4.7) | 25.9 (4.5)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 111.7 (11.3) | 113.4 (13.2) | 112.5 (12.3)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 76.2 (8.1) | 73.0 (10.6) | 74.6 (9.5)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 90.3 (7.0) | 91.5 (11.1) | 90.9 (9.2)
Total cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 184 [162 to 222] | 197 [171 to 215] | 194.5 [165 to 219]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 190 [131 to 228] | 142 [119 to 206] | 173 [126 to 214]
HDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 45 [38 to 52] | 46 [38 to 52] | 46 [38 to 52]
LDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 102 [82 to 131] | 109.7 [99.9 to 122.5] | 107 [88 to 123]
VLDL cholesterol [Median (Inter-Quartile Range); unit: mg/dL] | 37 [27 to 44] | 29 [25 to 45] | 33 [25.9 to 44.5]
Time in HAART [Median (Inter-Quartile Range); unit: months] | 36 [27 to 82] | 48 [25 to 100] | 45.5 [27 to 84]
Alanine aminotransferase [Median (Inter-Quartile Range); unit: UI/L] | 36 [28 to 46] | 35.5 [28 to 48] | 36 [28 to 46]
Aspartate aminotransferase [Median (Inter-Quartile Range); unit: UI/L] | 31 [24 to 36] | 28 [21 to 37] | 30 [22 to 36]
Lipoperoxides [Median (Inter-Quartile Range); unit: nM/mg protein] | 1.94 [1.6 to 3.1] | 2.0 [1.6 to 2.8] | 2.0 [1.6 to 2.8]
Total-glutathione [Median (Inter-Quartile Range); unit: μM] | 6.5 [2.6 to 30.6] | 4.0 [0 to 26.4] | 5.2 [1.8 to 28.8]
Oxidized-glutathione [Median (Inter-Quartile Range); unit: μM] | 0.3 [0 to 11.9] | 0.1 [0 to 2.2] | 0.2 [0 to 2.6]
Reduced-glutathione [Median (Inter-Quartile Range); unit: μM] | 4.4 [0 to 28.8] | 2.5 [0 to 23.1] | 3.4 [0 to 26.8]
Nitric oxide catabolites [Mean (Standard Deviation); unit: μM/ml] | 36.8 (14.2) | 39.0 (13.2) | 37.9 (13.6)
CD4 [Median (Inter-Quartile Range); unit: cel/µL] | 473 [398 to 555] | 595 [421 to 765] | 488 [407 to 729]
CD8 [Median (Inter-Quartile Range); unit: cel/µL] | 985 [652 to 1082] | 1117 [742 to 1553] | 1017 [708 to 1553]

OUTCOME MEASURES:

1. Primary Outcome: Change on Malondialdehyde After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: nM/mg protein
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
nM/mg protein | -1.18 [-1.94 to -0.23] | -0.9 [-1.2 to -0.12]

2. Secondary Outcome: Change on Total Glutathion After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: µM
Groups:
- Omega 3 Fatty Acids: Patients who received omega 3 fatty acids, 2.4 g per day, requiring intake 2 capsules (600mg each one) in the morning and 2 in the night...
- Placebo: Patiemts who received placebo for 6 months
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
µM | 32.9 [18.9 to 72.2] | 40.5 [26.4 to 65.8]

3. Secondary Outcome: Change on Nitric Oxide After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (Standard Deviation); unit: µM/ml
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
µM/ml | -21.1 (14.6) | -22.6 (14.6)

4. Secondary Outcome: Change on Viral Load After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: copies/ml
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
copies/ml | -396 [-1170 to -377] | 90 [-258 to 440]

5. Secondary Outcome: Change on Oxidized- Glutathion After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: µM
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
µM | 1.1 [-2.0 to 14.8] | 15.0 [7.6 to 19.1]

6. Secondary Outcome: Change on Reduced- Glutathion After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: µM
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
µM | 38.1 [13.6 to 52.0] | 27.9 [13.5 to 56.9]

7. Secondary Outcome: Change on Alanine Aminotransferase After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: UI/L
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
UI/L | 4.0 [-4.0 to 14.0] | 5.0 [-4.2 to 17.1]

8. Secondary Outcome: Change on Aspartate Aminotransferase After Treatment With Omega 3 Acids for 6 Months Compared With Placebo in HIV Seropositive Patients
Time Frame: The difference of this value at 6 months in relation to baseline value
Measure: Mean (95% Confidence Interval); unit: UI/L
Arm/Group | Omega 3 Fatty Acids | Placebo
Number analyzed (Participants) | 29 | 28
UI/L | 1.0 [-3.0 to 3.0] | 3.0 [-2.0 to 5.0]

ADVERSE EVENTS:
Arm/Group | Omega 3 Fatty Acids | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 2/35 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega 3 Fatty Acids (N=35) | Placebo (N=35)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
dizzines (Nervous system disorders) | 1 (1) | 0 (0)
biliar colic in patiet with cholelithiasis (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No